CLINICAL TRIAL: NCT01723436
Title: Pilot Study of Repeated Decision Making in Surrogates
Brief Title: Effects of Repeated Decision Making Among Surrogates of Seriously Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Scott Halpern, Assistant Professor of Medicine, Epidemiology, Health Policy and Medical Ethics, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 816697
Record Dates: First submitted 2012-11-01; First posted 2012-11-07 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Chemotherapy
Keywords: Decision fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- DLST Only (No Intervention): Surrogates will complete the Stroop test then answer the hypothetical life sustaining therapy (LST)
- Contemplate only (Experimental): Surrogates will contemplate each of the 3 scenarios but not make any decisions, then complete the Stroop test and answer the hypothetical LST question
  Interventions: Other: Hypothetical scenarios and related decisions
- Decide with advice (Experimental): Surrogates will make decisions on 4 scenarios with physician advice, then complete the Stroop test and answer the hypothetical LST question. Within this arm, surrogates will receive two positive recommendations (i.e. to go ahead with the intervention) and two negative recommendations (i.e. to decline the intervention). These positive and negative recommendations will be randomly assigned upon study enrollment. With four hypothetical scenarios, there are six possible options for recommendation variations.
  Interventions: Other: Hypothetical scenarios and related decisions
- Decide without advice (Experimental): Surrogates will make decisions on 4 scenarios without physician advice, then complete the Stroop test and the hypothetical LST question.
  Interventions: Other: Hypothetical scenarios and related decisions

INTERVENTIONS:
Other: Hypothetical scenarios and related decisions — Surrogates are exposed to three hypothetical medical scenarios that require varying levels of decision making. We will be assessing how this experience alters their subsequent choice to forego life sustaining therapy.
  Arms: Contemplate only; Decide with advice; Decide without advice

SUMMARY:
Decision making capacity fatigues after repeated decisions similar to skeletal muscle. The result is decision fatigue, in which subsequent decisions are altered toward the status quo. Surrogates are at risk for decision fatigue yet it has not been studied. We propose a randomized study in the outpatient setting in surrogates and patients at high risk for needing to make complex decisions, in an effort to determine the impact of decision fatigue on surrogate self-control and subsequent choices.

DETAILED DESCRIPTION:
Just as skeletal muscle fatigues after repeated use, decision-making capacity fatigues when repeated choices are made. This phenomenon, in which people experience diminished concentration and willpower after repeated decision-making, is termed decision fatigue. People experiencing decision fatigue are more likely to bias subsequent choices toward the status quo. By choosing the status quo, the decision-maker reserves the option to make an alternate choice at a later time, thereby preserving possibilities. Patients and their surrogates often make complex medical decisions for which they may have little experience. Although clearly at high risk, decision fatigue has not been studied in this population. To elucidate these questions, we propose a four-arm study of surrogates and patients in a population at high risk for making complex decisions. Surrogates will be randomly assigned to varied levels of decision making effort to assess for the development of resultant decision fatigue and whether it alters subsequent decisions.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following diagnoses: aplastic anemia, multiple myeloma, myelodysplastic syndrome, acute myeloid leukemia, stage IIIB or IV lung cancer, mesothelioma and/or stage IIIB or IV gastrointestinal cancer (pancreatic, biliary, esophageal, gastric, hepatocellular, colon), stage IV melanoma.
* Patients must have at least one surrogate at their clinic visit who is willing to enroll with them as a pair to be included.
* Surrogates are eligible if an eligible patient identifies them as as a surrogate and both consent for the study.
* All participants must be over the age 18
* All participants must be fluent in English

Exclusion Criteria:

* Patients and surrogates will be excluded if they are illiterate or have a medical condition known to alter Stroop performance. These include individuals who are visually impaired such that they cannot read a computer screen, blind or colorblind, patients given sedating medications during their appointment and individuals with past medical history of cerebrovascular accident, transient ischemic attack (TIA), seizure disorder, dementia or traumatic head injury with loss of consciousness.
* Patients will be ineligible if they have either tracheostomy or are currently on hemodialysis as these would significantly alter responses to the mechanical ventilation hypothetical scenario and the hypothetical life sustaining therapy question.
* Surrogates and patients are ineligible if their paired participant is excluded for any of the above reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Stroop Test Score | Approximately 15 minutes
  Measurement of score will be done at the conclusion of instrument completion. The Stroop test is a standard measure of self control that requires three tasks. The last task is the most difficult where the participant must suppress the urge to read the word which is the easier task and instead say the color it is printed in. Standard scoring is the number correct in the Word trial minus the Color-Word trials. This data will be collected immediately following completion.

SECONDARY OUTCOMES:
Evidence of status quo bias | Approximately 10 minutes
  Evidence of status quo bias as assessed by hypothetical decision to limit life sustaining therapy or to continue treatment. To assess for status quo bias, we will use the following technique: after the initial four hypothetical questions and Stroop testing, participants will be asked a hypothetical question about life sustaining therapy (LST). In the question, continuing life sustaining therapy will be counted as maintaining the status quo. This is based on current norms in American health care where life sustaining therapy is continued until a patient or surrogate specifically request otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Scott D. Halpern, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center for Advanced Medicine at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Vohs KD, Baumeister RF, Schmeichel BJ, Twenge JM, Nelson NM, Tice DM. Making choices impairs subsequent self-control: a limited-resource account of decision making, self-regulation, and active initiative. J Pers Soc Psychol. 2008 May;94(5):883-98. doi: 10.1037/0022-3514.94.5.883. PMID 18444745